CLINICAL TRIAL: NCT05562999
Title: Deep Versus Moderate Neuromuscular Blockade During Total HIP Replacement Surgery to Improve POstoperative Quality of Recovery and Immune Function: a Randomized Controlled Study
Brief Title: Impact of Deep Neuromuscular Blockade During Total Hip Replacement Surgery on Postoperative Recovery and Immune Function
Acronym: HIPPO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL81931.091.22
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-10

CONDITIONS: Neuromuscular Blockade; Innate Inflammatory Response; Quality of Life; Postoperative Complications
MeSH Terms: conditions — Inflammation; Postoperative Complications | interventions — Rocuronium; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deep neuromuscular blockade (Experimental): Participant will receive deep neuromuscular blockade (PTC 1-2)
  Interventions: Drug: Rocuronium Bromide
- Moderate neuromuscular blockade (Active Comparator): Participant will receive moderate neuromuscular blockade (TOF 1-2)
  Interventions: Drug: Rocuronium Bromide

INTERVENTIONS:
Drug: Rocuronium Bromide — Moderate NMB (TOF 1-2)
  Other Names: Bridion
  Arms: Moderate neuromuscular blockade
Drug: Rocuronium Bromide — Deep NMB (PTC 1-2)
  Other Names: Bridion
  Arms: Deep neuromuscular blockade

SUMMARY:
Monocenter randomized controlled trial to compare the effect of deep neuromuscular blockade (NMB) versus moderate NMB during total hip replacement surgery on postoperative quality of recovery and innate immune function.

DETAILED DESCRIPTION:
Rationale: Neuromuscular blockade agents (NMB) may enable surgeons to optimize exposure during hip surgery. With an increasing depth of NMB, manipulation of muscles and adjunctive tissues may be easier, therefore reducing damage to muscles and adjunct tissues. Accumulating evidence exists that the use of deep NMB in laparoscopic surgery is associated with a better quality of recovery and lower pain scores. However, whether this accounts for open surgery is still unknown.

In addition, surgery is associated with postoperative immune suppression. Surgical stress and damage cause the release of Danger Associated Molecular Patterns (DAMPs). After trauma and sepsis, the release of DAMPs is associated with immune paralysis and a higher susceptibility to infectious complications. Previous research indicates that DAMPS are the origin of postoperative immune suppression. The use of deep NMB in hip surgery may reduce surgical damage and thereby lead to a better quality of recovery and secondarily a better preservation of immune cell function.

Primary objective: To establish the relationship between the use of deep neuromuscular blockade (NMB) versus moderate NMB and the quality of recovery after total hip replacement surgery (THR) Secondary objective: To establish the relationship between the use of deep NMB versus moderate NMB and innate immune function after THR surgery

Study design: A monocenter, blinded, randomized controlled clinical trial

Study population: adults who are scheduled for primary or secondary hip replacement surgery under general anaesthesia.

Intervention: Patients will be randomized between a deep NMB (post tetanic count (PTC) 1-2) and moderate NMB (Train-of-four (TOF) 1-2)

Primary endpoint: Quality of Recovery score (QoR-40) at postoperative day 1.

Secondary endpoints: postoperative innate immune function, QoR-40 at postoperative day 30, 30-day postoperative (infectious) complications, postoperative pain scores and opioid consumption

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Scheduled for total hip replacement surgery under general anaesthesia
* Informed consent obtained

Exclusion Criteria:

* Insufficient control of the Dutch language to read the patient information and to fill out de questionnaires
* Known or suspected hypersensitivity to rocuronium or sugammadex
* Deficiency of vitamin K dependent clotting factors or coagulopathy
* Severe renal disease (creatinine clearance <30 ml/min), including patients on dialysis
* Severe liver disease (Child-Pugh Classification C)
* Known or suspected neuromuscular disorders impairing neuromuscular function
* Women who are or may be pregnant or currently breastfeeding
* Chronic use of psychotropic drugs
* Use of immunomodulatory medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery 40 (QoR-40) questionnaire score | Postoperative day 1
  40 points (minimum: extremely poor quality of recovery) to 200 points (maximum: excellent quality of recovery)

SECONDARY OUTCOMES:
Quality of Recovery 40 (QoR-40) questionnaire score | Postoperative day 30
  40 points (minimum: extremely poor quality of recovery) to 200 points (maximum: excellent quality of recovery)
Immune function represented by serum cytokine | Postoperative day 1
  Serum cytokine IL-6 level
Immune function represented by IL-10 | Postoperative day 1
  Serum cytokine IL-10 level
Immune function represented by TNF-a | Postoperative day 1
  Serum cytokine TNF-a level
Immune function represented by ex-vivo IL-6 production capacity | Postoperative day 1
  Ex-vivo IL-6 production capacity upon whole blood Lipopolysaccharide(LPS) stimulation
Immune function represented by ex-vivo IL-10 production capacity | Postoperative day 1
  Ex-vivo IL-10 production capacity upon whole blood LPS stimulation
Pain score by numeric pain rating (NRS) scale | During hospital admission up to 3 days postoperative
  pain scores with NRS 0 (no pain) to 10 (severe pain)
Postoperative complications | 30 postoperative days
  postoperative complications scored by Clavien-Dindo classification; grade 0 (no deviation from ideal) grade 5 (death of patient)
Infectious postoperative complications | 30 postoperative days
  Postoperative infectious complications scored the definitions of the StEP-COMPAC group initiative
Analgesia consumption | During hospital admission up to 3 days postoperative
  non-cumulative and cumulative opioid use per day in morphine equivalent

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
All data will be analyzed for publication. After that it belongs to Radboud umc where other researchers of Radboud umc may or may not include this database to their study. But there will be no active sharing

REFERENCES:
- [Derived] Jacobs LMC, Bijkerk V, van Eijk LT, Joosten LAB, Keijzer C, Visser J, Warle MC. The effect of general versus spinal anesthesia on perioperative innate immune function in patients undergoing total hip arthroplasty. BMC Anesthesiol. 2025 Jan 7;25(1):10. doi: 10.1186/s12871-024-02883-1. PMID 39773137
- [Derived] Bijkerk V, Visser J, Jacobs LMC, Keijzer C, Warle MC. Deep versus moderate neuromuscular blockade during total hip arthroplasty to improve postoperative quality of recovery and immune function: protocol for a randomised controlled study. BMJ Open. 2023 Aug 28;13(8):e073537. doi: 10.1136/bmjopen-2023-073537. PMID 37640469